CLINICAL TRIAL: NCT05906875
Title: A Novel Balance Program to Improve Balance in People With Parkinson's Disease: A Feasibility Study
Brief Title: A Novel Balance Program to Improve Balance in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Collaborators: The Touro College and University System (Other)
Responsible Party: Principal Investigator, Michael Tautonico, Assistant Professor, New York Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS- IRB
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-12

CONDITIONS: Rehabilitation Exercise; Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prove feasible to integrate into an existing community group exercise program (Other): Prove feasible to integrate into an existing community group exercise program and Decrease the number of fall risk factors
  Interventions: Other: Lateral Stepping Exercise 1; Other: Lateral Stepping Exercise 2; Other: Lateral Stepping Exercise 3; Other: Lateral Stepping Exercise 4; Other: Lateral Stepping Exercise 5

INTERVENTIONS:
Other: Lateral Stepping Exercise 1 — 1. Standing hip abduction: Performed without and with resistance bands and/or support. The participant will raise one leg out to the side and return. If using a resistance band, one end of the band will be secured to a stable surface and the other end placed around one of the participants' ankles. The banded leg will be raised to the side. Three sets of 8-12 repetitions will be performed per side.
Other: Lateral Stepping Exercise 2 — 2. Lateral stepping: Performed without and with resistance bands. The participant will perform a series of steps to the side. If using a resistance band, the band will be placed around both ankles in a 'loop' and the participant will perform the lateral stepping. Three sets of 8-12 repetitions will be performed per side per subject.
Other: Lateral Stepping Exercise 3 — 3. Single leg stance: The participant will stand on one leg with support as needed. The contralateral knee will be held at 45 degrees throughout the exercise. The instructor will observe to ensure the bent leg does not contact the ground. Three repetitions of static stance per side will be performed with a goal of 30 seconds, and a maximum time of 60 seconds, per repetition.
Other: Lateral Stepping Exercise 4 — 4. Staggered stance mini-squat: Participants will stand with the feet hip-width apart and one leg placed a short step forward. The participant will squat straight down keeping the trunk upright and return to an upright position.
Other: Lateral Stepping Exercise 5 — 5. Lateral Reactive Postural Control: The participant will lean into the researcher's hand to shift their center of mass outside of their base of support. Hand placement will be at the glenohumeral joint and the pelvis. The researcher will withdraw support and guard the participant as the participant regains their balance. This is item 6 on the Mini-BESTest assessment that will be incorporated as an intervention. To be performed 3x per side.

SUMMARY:
The purpose of this exploratory single-blinded feasibility study is to explore the effects of a lateral stepping program integrated into an existing community-based group exercise program for people with PD. The researchers hypothesize that participation in a lateral stepping program a minimum of 2 times/week for 8 weeks, in addition to RSB class participation is feasible in middle to late stage PD and will decrease fall risk factors. The researchers also hypothesize that the integration of this program into an existing community-based RSB program will be deemed feasible as shown by the number of sessions attended by each participant.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of idiopathic PD stages II, III, or IV of the Hoehn and Yahr scale
2. 50-85 years inclusive
3. Subjects must be enrolled in RSB at NY Tech and attend at least 1 day per week for a minimum of 4 weeks prior to the first baseline assessment
4. English speaking.
5. Stable PD medication regime.

Exclusion Criteria:

1. Any cardiovascular or other medical condition that would affect participation
2. Any hip and/or knee surgery or other injury that would prevent full participation in the intervention
3. Neurological conditions other than PD
4. Montreal Cognitive Assessment of ≤21
5. Pain that interferes with testing 13
6. Current participation in other strengthening, stretching or balance programs other than Rock Steady Boxing at NY Tech
7. Inability to understand and fully participate in this study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
The Mini-BESTest | 10-15 minutes
  Performance measure, validated in people with PD, aimed to target and identify 6 different balance control systems
The Functional Gait Assessment | 5-20 minutes
  Validated for people with PD is a performance measure validated in people with PD that is used to assess balance in the higher-functioning older adult and examines ambulation and the ability to perform motor tasks while ambulating
The Multidirectional Functional Reach Test | Less than 5 minutes
  Used to assess stability when displacing a person's balance in a forward, lateral, and backward direction
The Four-Square Step Test | less than 5 minutes
  Validated for people with PD is used to measure a patient's fall risk. The test requires a stopwatch and 4 canes laid in a cross pattern. The canes crossed pattern makeup 4 quadrants; quadrant 1 (bottom left), quadrant 2 (top left), quadrant 3 (top right), and quadrant 4 (bottom right). The subject is timed while they step clockwise, and then counterclockwise throughout the quadrants. An assistive device may be used.
The Activities Balance Confidence Scale | 5-10 minutes
  Validated for people with PD, is a self-report measure of balance confidence while performing various common activities. Scale is from 0% to 100% with 100% being the most confident in their balance in a criterion.
The Parkinson's Disease Questionnaire-39 | approximately 10 minutes
  39-item self-administered questionnaire designed to assess 8 different quality-of-life domains. Uses a 5-point ordinal scale with 0 being never and 5 being always. Lower scores indicate a lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States